CLINICAL TRIAL: NCT06263205
Title: Clinical Investigation of Wound Management Following Gastrointestinal Tumor Surgery: Comparing Outcomes of Dressing Changes Versus Non-Dressing Techniques
Brief Title: Wound Management Following Gl Tumor Surgery: Comparing Outcomes of Dressing Changes Versus Non-Dressing Techniques
Acronym: Dressing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Shanghai Changzheng Hospital (Other); Changhai Hospital (Other); Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dressing
Record Dates: First submitted 2024-01-15; First posted 2024-02-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Tumors; Surgical Wound Infection; Pain, Postoperative
MeSH Terms: conditions — Digestive System Neoplasms; Surgical Wound Infection; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Dressing Group (Experimental): Participants in this group will receive standard wound disinfection and dressing immediately after gastrointestinal tumor surgery. At 48 hours post-surgery, the dressing will be removed and the wound will be left exposed without any disinfection or reapplication of dressing. This state will be maintained until suture removal at 7-14 days postoperatively. This arm aims to evaluate the outcomes when the surgical wound is kept exposed, in contrast to traditional dressing methods.
  Interventions: Procedure: Non-Dressing of Surgical Wound
- Dressing Group (Active Comparator): Participants in this group will receive standard postoperative care. Their surgical wounds will be covered with dressings immediately after surgery, and these dressings will be changed every 48 hours (including disinfection and reapplication of dressing) until suture removal at 7-14 days postoperatively. This group serves as the comparator for assessing the non-dressing approach.
  Interventions: Procedure: Regular Dressing Change of Surgical Wound

INTERVENTIONS:
Procedure: Non-Dressing of Surgical Wound — Participants will receive standard wound disinfection and dressing immediately after surgery. Unlike traditional methods, the dressing will be removed at 48 hours post-surgery, and the wound will then be left exposed without disinfection or coverage** until suture removal (7-14 days postoperatively). This method evaluates the effects of wound exposure on healing, pain, and healthcare costs.
  Arms: Non-Dressing Group
Procedure: Regular Dressing Change of Surgical Wound — This intervention involves standard postoperative wound care. After surgery, wounds will be disinfected and covered with dressings. Dressings will be changed every 48 hours (with disinfection and reapplication) until suture removal (7-14 days postoperatively), following traditional wound management practices.
  Arms: Dressing Group

SUMMARY:
The goal of this clinical trial is to assess the effectiveness and safety of non-dressing (exposed wound) versus dressing techniques in postoperative wound management for patients with gastrointestinal tumors. The main questions it aims to answer are:

1. Does non-dressing of postoperative wounds in gastrointestinal tumor surgery provide equivalent or better wound healing compared to traditional dressing techniques?
2. Can non-dressing of postoperative wounds reduce patient pain and healthcare costs? Participants in this study, who are diagnosed with gastrointestinal tumors and undergoing surgery, will be randomly assigned to either the non-dressing group or the dressing group. The non-dressing group will have their surgical wounds left exposed after initial postoperative care, while the dressing group will receive regular wound dressing changes every 48-72 hours. Researchers will compare these two groups to see if there are differences in the rate of wound complications, pain levels, and overall healthcare costs.

This study aims to provide evidence-based recommendations for postoperative wound care in gastrointestinal tumor surgeries, potentially improving patient outcomes and reducing medical expenses.

DETAILED DESCRIPTION:
Research Objectives and Design:

This study is a prospective, randomized controlled trial primarily aimed at comparing the efficacy of wound healing between non-dressing and dressing methods post-gastrointestinal tumor surgery. The secondary objective is to evaluate the effectiveness of the non-dressing approach in reducing postoperative pain and medical expenses.

Inclusion Criteria and Sample Size:

The study plans to enroll 212 patients aged 75 years or younger, diagnosed pathologically with gastrointestinal tumors and scheduled for curative surgery or open gastrointestinal bypass surgery. Participants must have an ECOG (Eastern Cooperative Oncology Group) performance status score of 0/1 and be capable of understanding and signing the informed consent. Exclusion criteria include inability to complete postoperative follow-up, ineligibility for surgical treatment, concurrent skin diseases, history of abdominal trauma or surgery, other uncontrolled severe diseases, ongoing other cancer treatments, and current use of drugs that may affect wound healing.

Study Methodology:

Participants will be randomly assigned to one of two groups: a non-dressing group (Group A) and a dressing group (Group B). Group A will have dressings removed 48 hours post-surgery and keep the wound exposed unless signs of infection are present. Group B will undergo regular dressing changes every 48 to 72 hours until sutures are removed between the 7th and 14th postoperative days. Both groups will be closely monitored for wound treatment and complications such as fat liquefaction, infection, and wound dehiscence.

Withdrawal/Early Termination Criteria:

Patients may withdraw from the study voluntarily at any time. Researchers can also decide to withdraw a patient if continued treatment is deemed not in the patient's best interest. Reasons for withdrawal include but are not limited to other concurrent diseases, death, relapse, complications, receiving non-study treatments, or patient's request to exit the study.

Follow-up Plan:

The study will conduct stringent follow-ups, including observation and assessment of the surgical wound 30 days post-surgery, recording the frequency of dressing changes, total costs, pain scores, and wound comfort levels. The follow-up endpoints include patient withdrawal, change in treatment modality, disease progression, death, or reaching the study's end date.

Observation and Evaluation during the Trial:

All trial procedures must be preceded by obtaining informed consent approved by an ethical committee. All data collected during the trial will be statistically analyzed following the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≤ 75 years.
2. Scheduled to undergo gastrointestinal surgery for gastrointestinal cancer (pathologically confirmed).
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
4. Possesses sufficient cognitive ability to understand the study protocol and voluntarily signs a written informed consent form.

Exclusion Criteria:

1. Presence of significant barriers to completing postoperative follow-up (e.g., severe sensory/cognitive impairment, inability to adhere to follow-up plan, lack of reliable contact methods, residence >6 hours from study center).
2. Concurrent active skin diseases that may affect wound healing (e.g., psoriasis, chronic eczema, atopic dermatitis) located at or near the surgical incision site.
3. History of major abdominal trauma or prior abdominal surgery resulting in abdominal wall deformity or extensive scarring that may affect incision healing or assessment.
4. Current diagnosis of any other uncontrolled severe comorbid conditions (e.g., uncontrolled other malignant tumors, acute or persistent chronic infections) that may pose additional risks or confound study outcomes.
5. Planned or ongoing receipt of any other anticancer treatments (chemotherapy, targeted therapy, biological therapy, radiotherapy) or long-term immunosuppressive therapy during the perioperative period.
6. Current long-term or high-dose use of systemic corticosteroids or any other medications that may significantly affect wound healing (topical/inhaled/low-dose steroids allowed if assessed by investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1138 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite wound complications within 30 days after surgery | Within 30 days after surgery
  This is a composite endpoint including surgical site infection, wound dehiscence, hematoma/seroma requiring intervention, fat liquefaction, and delayed wound healing. The non-inferiority of the "no dressing change" strategy versus the "routine dressing change" strategy will be tested using the Farrington-Manning test. The pre-specified non-inferiority margin (Δ) is 6%. Non-inferiority will be established if the upper limit of the two-sided 95% confidence interval for the difference in incidence rates (no dressing change minus routine dressing change) is below 6%.
  Time Frame: Up to 30 days after surgery.

SECONDARY OUTCOMES:
Patient Pain Levels | Pain scores will be assessed at three specific time points during the early postoperative period: on postoperative day 2, day 4, and day 6. The primary comparison will be the trend of pain scores across these time points between the two groups.
  Postoperative incisional pain intensity will be assessed using the Visual Analog Scale (VAS). The VAS is a validated, self-reported tool consisting of a 10-cm horizontal line anchored by two verbal descriptors: "0 = No pain" on the left end and "10 = Worst imaginable pain" on the right end. Participants will be instructed to mark a point on the line that best represents their current pain intensity at rest. The distance from the left anchor to the mark is measured in centimeters, yielding a pain score ranging from 0 to 10, with higher scores indicating greater pain intensity.
  To minimize assessment bias, pain evaluations will be conducted by research staff who are trained in standardized administration and are blinded to the treatment group assignment (where feasible) during follow-up assessments. The assessments will be performed at predefined time points postoperatively.
Medical Costs Associated with Wound Care | From the time of surgery up to 30 days post-surgery
  This measure evaluates the total medical costs associated with wound care following surgery. This includes the costs of dressings and the frequency of dressing changes. The aim is to compare these costs between the non-dressing and dressing groups to determine if non-dressing can help reduce healthcare expenses.

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Xu, MD, PhD, Principal Investigator — Fudan University
Locations (4):
- China (4):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Changzheng Hospital, Navy Medical University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, School of Medicine, Tongji University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Naval Medical University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
The IPD that will be shared includes de-identified participant data encompassing demographic information, clinical data, and outcomes of interventions (dressing changes vs. non-dressing techniques). This may also include study protocol, statistical analysis plan, and informed consent form. All shared data will be de-identified to protect participant privacy and confidentiality. Researchers accessing the data will be required to sign a data access agreement that includes a commitment to using the data only for research purposes and not attempting to identify individual participants.
Supporting Information: SAP
Time Frame: The IPD will be available for sharing 12 months after the publication of the main study results and will remain accessible for five years.
Access Criteria: Data access will be granted to researchers who provide a methodologically sound proposal, which will be reviewed and approved by an independent review committee. The proposal must be approved by an ethics committee or institutional review board.

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Kim HH, Han SU, Kim MC, Hyung WJ, Kim W, Lee HJ, Ryu SW, Cho GS, Song KY, Ryu SY. Long-term results of laparoscopic gastrectomy for gastric cancer: a large-scale case-control and case-matched Korean multicenter study. J Clin Oncol. 2014 Mar 1;32(7):627-33. doi: 10.1200/JCO.2013.48.8551. Epub 2014 Jan 27. PMID 24470012
- [Result] Hyung WJ, Yang HK, Han SU, Lee YJ, Park JM, Kim JJ, Kwon OK, Kong SH, Kim HI, Lee HJ, Kim W, Ryu SW, Jin SH, Oh SJ, Ryu KW, Kim MC, Ahn HS, Park YK, Kim YH, Hwang SH, Kim JW, Cho GS. A feasibility study of laparoscopic total gastrectomy for clinical stage I gastric cancer: a prospective multi-center phase II clinical trial, KLASS 03. Gastric Cancer. 2019 Jan;22(1):214-222. doi: 10.1007/s10120-018-0864-4. Epub 2018 Aug 20. PMID 30128720
- [Result] Ushiku H, Hosoda K, Yamashita K, Katada N, Kikuchi S, Tsuruta H, Watanabe M. A Risk Model for Surgical Site Infection in the Gastric Cancer Surgery Using Data of 790 Patients. Dig Surg. 2015;32(6):472-9. doi: 10.1159/000440703. Epub 2015 Oct 28. PMID 26505458
- [Result] Inokuchi M, Sugita H, Otsuki S, Sato Y, Nakagawa M, Kojima K. Laparoscopic distal gastrectomy reduced surgical site infection as compared with open distal gastrectomy for gastric cancer in a meta-analysis of both randomized controlled and case-controlled studies. Int J Surg. 2015 Mar;15:61-7. doi: 10.1016/j.ijsu.2015.01.030. Epub 2015 Jan 31. PMID 25644544
- [Result] Nichols RL. Preventing surgical site infections: a surgeon's perspective. Emerg Infect Dis. 2001 Mar-Apr;7(2):220-4. doi: 10.3201/eid0702.010214. PMID 11294711
- [Result] Chetter IC, Oswald AV, Fletcher M, Dumville JC, Cullum NA. A survey of patients with surgical wounds healing by secondary intention; an assessment of prevalence, aetiology, duration and management. J Tissue Viability. 2017 May;26(2):103-107. doi: 10.1016/j.jtv.2016.12.004. Epub 2016 Dec 21. PMID 28049612
- [Result] Giaquinto-Cilliers MGC, Nair A, Von Pressentin KB, Coetzee F, Saeed H. A 'game of dressings': Strategies for wound management in primary health care. S Afr Fam Pract (2004). 2022 Feb 28;64(1):e1-e8. doi: 10.4102/safp.v64i1.5462. PMID 35261259
- [Result] Upton D, Solowiej K. The impact of atraumatic vs conventional dressings on pain and stress. J Wound Care. 2012 May;21(5):209-15. doi: 10.12968/jowc.2012.21.5.209. PMID 22584737
- [Result] Heal C, Buettner P, Raasch B, Browning S, Graham D, Bidgood R, Campbell M, Cruikshank R. Can sutures get wet? Prospective randomised controlled trial of wound management in general practice. BMJ. 2006 May 6;332(7549):1053-6. doi: 10.1136/bmj.38800.628704.AE. Epub 2006 Apr 24. PMID 16636023
- [Result] Dumville JC, Gray TA, Walter CJ, Sharp CA, Page T, Macefield R, Blencowe N, Milne TK, Reeves BC, Blazeby J. Dressings for the prevention of surgical site infection. Cochrane Database Syst Rev. 2016 Dec 20;12(12):CD003091. doi: 10.1002/14651858.CD003091.pub4. PMID 27996083
- [Result] Law NW, Ellis H. Exposure of the wound--a safe economy in the NHS. Postgrad Med J. 1987 Jan;63(735):27-8. doi: 10.1136/pgmj.63.735.27. No abstract available. PMID 3671224
- [Result] Furka A, Simko C, Kostyal L, Szabo I, Valikovics A, Fekete G, Tornyi I, Oross E, Revesz J. Treatment Algorithm for Cancerous Wounds: A Systematic Review. Cancers (Basel). 2022 Feb 25;14(5):1203. doi: 10.3390/cancers14051203. PMID 35267512